CLINICAL TRIAL: NCT01487954
Title: Alkaline Water Consumption to Reduce Skin Radiation Toxicity in Women With Breast Cancer
Brief Title: Alkaline Water in Reducing Skin Toxicity in Women With Breast Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CASE2109; NCI-2010-01233 (Other: NCI/CTRP)
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Radiation Toxicity; Recurrent Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
Keywords: skin reactions secondary to radiation therapy
MeSH Terms: conditions — Radiation Injuries; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: alkaline water (Experimental): Patients undergo external beam radiation therapy QD, 5 days a week for 6 weeks. Patients drink 8 ounces of alkaline water within 30 minutes immediately prior to and after undergoing radiation therapy.
  Interventions: Dietary Supplement: alkaline water; Radiation: external beam radiation therapy (EBRT)
- Arm II: distilled water (Active Comparator): Patients undergo external beam radiation therapy as in arm I. Patients also drink 8 ounces of distilled water within 30 minutes immediately prior to and after undergoing radiation therapy
  Interventions: Dietary Supplement: distilled water; Radiation: external beam radiation therapy (EBRT)

INTERVENTIONS:
Dietary Supplement: alkaline water — Patients drink 8 ounces of alkaline water within 30 minutes immediately prior to and after undergoing radiation therapy.
  Arms: Arm I: alkaline water
Dietary Supplement: distilled water — Patients also drink 8 ounces of distilled water within 30 minutes immediately prior to and after undergoing radiation therapy.
  Arms: Arm II: distilled water
Radiation: external beam radiation therapy (EBRT) — Patients undergo external beam radiation therapy QD, 5 days a week for 6 weeks.

SUMMARY:
This phase II trial is studying how well alkaline water works in reducing skin toxicity in women with breast cancer undergoing radiation therapy. Alkaline water may reduce radiation therapy-related skin toxicity in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. The goal of this two-phase study is to assess the rate of grade 2 or higher radiation-related skin toxicity in adult patients with breast malignancies after administration of alkaline (pH 9.0) or distilled (pH 7.0) water consumed immediately prior to and after daily radiation treatments.

OUTLINE:

FEASIBILITY PHASE: Patients undergo external beam radiation therapy once daily (QD), 5 days a week for 6 weeks. Patients drink 8 ounces of alkaline water within 30 minutes immediately prior to and after undergoing radiation therapy.

INTERVENTION PHASE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo external beam radiation therapy QD, 5 days a week for 6 weeks. Patients drink 8 ounces of alkaline water within 30 minutes immediately prior to and after undergoing radiation therapy.

ARM II: Patients undergo external beam radiation therapy as in arm I. Patients also drink 8 ounces of distilled water within 30 minutes immediately prior to and after undergoing radiation therapy.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage 0-IV breast cancer and have a treatment plan consisting of 62Gy (31 fractions) of total breast radiation therapy to be eligible; patients are eligible if they have received any number of prior chemotherapies; patients having received chemotherapy prior to radiation will be stratified among randomization groups during the second phase of this study
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients receiving any investigational chemotherapeutic agents during planned radiation or any prior breast or chest wall radiation treatments are excluded
* Patients receiving concurrent chemotherapy are excluded because of an increased relative risk of skin toxicity; patients taking daily proton-pump inhibitor or H2-blocker antacid medications are excluded because of predicted interference of alkaline water consumption and stomach pH; herceptin for the purposes of this clinical trial would be considered a chemotherapy, and as such, patients receiving herceptin chemotherapy during radiation would not be eligible for participation in this protocol
* Patients with a history of any prior malignancy except non-melanoma skin cancer or carcinoma in-situ of the cervix not in remission for twelve months are excluded; patients with known brain metastases are excluded from this clinical trial because of their overall poor prognosis
* Pregnancy excludes female patients from this study because radiation is potentially teratogenic and abortifacient; screening beta-hcg levels and clinically-indicated diagnostic tests will be used to determine eligibility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals-Westlake, Westlake, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Alkaline Water | Arm II: Distilled Water
Started | 29 | 16
Safety lead-in | 10 | 0 (Only the first 10 patients in the alkaline group were analyzed, as that was the experimental group.)
Completed | 29 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Alkaline Water | Arm II: Distilled Water | Total
Number analyzed (Participants) | 29 | 16 | 45
Age, Continuous [Median (Full Range); unit: years] | 57 [45 to 79] | 53 [40 to 66] | 57 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 16 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 16 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 16 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Acute and Grade 2 or Higher Radiation-related Skin Toxicity as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Information will include the type, severity, time of onset and resolution of its onset, and its probable association with the study regimen. Frequency tables will be constructed to summarize observed incidents by severity and type of toxicity during weekly radiation treatment and 1 month after radiation treatment. Observed toxicity differences among the treatment arms may be reported in frequency tables.
Time Frame: at 1 month after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Alkaline Water | Arm II: Distilled Water
Number analyzed (Participants) | 29 | 16
percentage of participants | 38 | 38

2. Secondary Outcome: Change in Urine pH
Description: A paired sample t-test (a=0.05) assessing change in urine pH between before treatment day 0 and after radiation and alkaline water treatment day 33.
Time Frame: at baseline and at week 5 (day 33)
Population: Only the first ten patients in the alkaline water group, who took part in the safety lead-in portion of the study were analyzed for urine pH
Measure: Mean (Standard Deviation); unit: units on pH scale
Arm/Group | Arm I: Alkaline Water | Arm II: Distilled Water
Number analyzed (Participants) | 10 | 0
units on pH scale
  pH at baseline | 5.6 (0.7) |
  pH at day 33 of treatment | 6.1 (1.0) |

ADVERSE EVENTS:
Time Frame: 30 days after treatment
Arm/Group | Arm I: Alkaline Water | Arm II: Distilled Water
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/16
Other Adverse Events (participants affected / at risk) | 26/29 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Alkaline Water (N=29) | Arm II: Distilled Water (N=16)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Increased blood level of a liver enzyme (ALT/SGPT)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) — Increased blood level of a liver enzyme (AST/SGOT)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Chest wall pain
Skin infection (Infections and infestations) | 0 (0) | 1 (1) — cellulitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Alkaline Water (N=29) | Arm II: Distilled Water (N=16)
dermatitis (Skin and subcutaneous tissue disorders) | 26 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes